CLINICAL TRIAL: NCT02127450
Title: Carbapenem-resistant Enterobacteriaceae: Prevalence, Risk Factors and Impact of the Use of the Phenotypic Algorithm for the Detection of Carbapenemases
Acronym: E-CARB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 12025
Record Dates: First submitted 2014-04-16; First posted 2014-04-30 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Enterobacteria Non Susceptible to Carbapenem Carrier; Enterobacteria Susceptible to Carbapenem Carrier
Keywords: Enterobacteriaceae; non-susceptible to carbapenem; carbapenemases; prevalence; screening algorithm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Enterobacteriaceae Isolates non-susceptible to carbapenem (NS -CARB)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Case: NS-CARB positive: Patient with a clinical sample positive for a NS-CARB Enterobacteriaceae
- Control 1: non-NS-CARB positive: Patient with clinical sample positive for a non-NS-CARB Enterobacteriaceae
- Control 2 : negative sample: Patient having had clinical sample(s) being stayed negative since the beginning of his admission and up to 3 days after the detection of the case

SUMMARY:
The non-susceptibility of enterobacteriaceae isolates to carbapenem (CARBA) is an emerging concern with a high impact on infectious disease therapy. carbapenemase (CARBase) production are one of the mechanisms of resistance to CARBA. When CARBase production is suspected or proved, specific hygiene measures have to be applied in any hospital. Detecting CARBase in the routine in any laboratory is difficult. it will be useful to standardize them detection to control the emergence.

DETAILED DESCRIPTION:
The non-susceptibility of enterobacteriaceae isolates to carbapenem (CARBA) is an emerging concern with a high impact on infectious disease therapy because CARBA are often the alone antibiotics available to cure severe infections due to extended-spectrum β-lactamase (ESBL)-producing isolates. Two mechanisms of resistance to CARBA have been identified: membrane impermeability associated with ESBL or cephalosporinase production and carbapenemase (CARBase) production. When CARBase production is suspected or proved, specific hygiene measures have to be applied in any hospital in order to avoid the dissemination of the CARBase-producing strain and insure patient safety. Prevalence rate of non-susceptible (NS) isolates to CARB, the proportion of the two types of mechanisms of resistance to CARB and the factors associated with CARB- NS isolates are still unknown in France. Moreover, detecting CARBase in the routine in any laboratory is difficult. Providing data regarding all of these points will be useful for any hospital and will permit to optimize the management of the patients suspected or proved to harbor a CARBase-producing Enterobacteriaceae isolate.

ELIGIBILITY:
Inclusion Criteria:

* Case: Patient with a clinical sample positive for a NS-CARB Enterobacteriaceae
* Control 1: Patient with clinical sample positive for a non-NS-CARB Enterobacteriaceae and hospitalised in the same type of ward as that case
* Control 2: Patient having had clinical sample(s) being stayed negative since the beginning of his admission and up to 3 days after the detection of the case, hospitalised in any type of ward in the hospital

Exclusion Criteria:

* the patient with digestive ER-CARB

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patient hospitalised for more than 24 hours , with a clinical sample positive for a NS-CARB Enterobacteriaceae
  * Patient hospitalised for more than 24 hours with clinical sample positive for a non-NS-CARB Enterobacteriaceae and hospitalised in the same type of ward as that case
  * Patient hospitalised for more than 24 hours having had clinical sample(s) being stayed negative since the beginning of his admission and up to 3 days after the detection of the case, hospitalised in any type of ward in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rate of CARB-NS isolates and among them the proportion of those producing CARBase. | 1 year
  Determining the prevalence rate of CARB-NS isolates and among them the proportion of those producing CARBase for all enterobacterial species and for each species. CARBase production will be determined by using in a phenotypic algorithm previously established on the basis on commercialized tests and by molecular methods.
  Determining by using a prospective case-control-control study the factors associated with a clinical sample positive for a NS-CARB isolate by distinguishing isolates non-CARBase-producing and isolates CARBase-producing.This study will be carried out during one year in 18 hospitals across France whose laboratory will participate in the prevalence study. The variables independently associated with a clinical sample positive for either a NS-CARB, non-CARBase-producing isolate or a NS-CARB, CARBase-producing isolate will be determined in a multivariate analysis.

SECONDARY OUTCOMES:
Detection of CARBase producing isolates as a measure of the diagnostic value of the phenotypic algorithm | 1 year
  Assessing the diagnostic value (sensitivity, specificity, positive predictive value and negative predictive value) of the phenotypic algorithm for the detection CARBase producing isolates by using the molecular methods as Gold standard method
Impact of the use of the phenotypic algorithm on the management of the patients identified as carrier of NS-CARB isolate. | 1 year
  Assessing the impact of the use of the phenotypic algorithm on the management of the patients identified as carrier of NS-CARB isolate (case) in the 18 hospitals : (i) time between the period at which the isolate is identified as NS-CARB and, on the one hand, knowledge acquisition by the Hygiene team and the medical staff of the presence of the case, and on the other hand, the period at which barrier precautions are implemented by distinguishing the type of barrier precautions implemented (standard or with dedicated non-medical staff) (ii) the duration of the implementation of barrier precaution with regard to the results concerning the production or the non-production of a CARBase by the NS-CARB isolate . The results of this study will be compared with the results obtained during a previous study in which the phenotypic algorithm had not been used.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Nicolas-Chanoine, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided